CLINICAL TRIAL: NCT06497205
Title: AMBulatory Fetal ECG Monitoring in Low and High-Risk Pregnancies
Status: Recruiting | Type: Observational
Sponsor: Biorithm Pte Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: AMBER2
Record Dates: First submitted 2024-07-04; First posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Pregnancy Related

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control Group: low risk ASPRE
- FGR Group: FGR according to definition of ISUOG
- Diabetic Group: insulin dependent diabetes

SUMMARY:
This study is a planned research project to test and demonstrate the feasibility of using the Femom device for monitoring fetal heart rate remotely.

The main goal is to learn if the remote recordings using Femom provide reliable information about the baby's heart rate. We will also establish reference standards of heart rate variability in uncomplicated pregnancies at different stages of pregnancy. Additionally, we will compare the heart rate variability in FGR and diabetic pregnancies to normal pregnancies.

DETAILED DESCRIPTION:
The Femom device is a non-invasive fetal ECG (NIFECG) device which has been developed for self application and remote monitoring. Women from three different cohort groups (controls, FGR and insulin dependent diabetes) will be approached and asked to monitor their baby at home once a day. Women in the control group will be asked to do this once a day for one week, the FGR pregnancies until delivery and the insulin dependent diabetics just from 36 weeks until delivery.

The data will be collected and analysed retrospectively to assess compliance of the participants with the study protocol, signal quality and establish reference standards in relation to gestation within the control group. Heart rate variability measures in the FGR and diabetes arm will be compared to the reference standards in the control group. Outcomes of the pregnancy.

Feedback regarding the usability of the device will also be collected using a feedback questionnaire to assess the feasibility of home antenatal monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Singleton live pregnancy
* > 26 weeks gestational age
* Able to speak English or available NHS interpreter

Exclusion Criteria:

* Women below 18 years of age
* Women with an intellectual or mental impairment
* Women with a known allergy or hypersensitivity to ECG gel electrodes
* Known fetal cardiac or genetic abnormality.
* Patient with existing dependent or unequal relationships with any member of the research team, the researchers(s) and/or the person undertaking the recruitment/consent process.
* Inability to access interpreter.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women booked for antenatal care at St. George's hospital or women under the care of the Fetal medicine unit at St. George's hospital will be invited to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2024-03-19 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
FHR | 60 minutes
  FHR agreement between Femom system and standard of care (CTG)
MHR | 60 minutes
  MHR agreement between Femom system and standard of care (CTG)

CONTACTS AND LOCATIONS:
Overall Officials: Amarnath Bhide, MBBS, PHD, Principal Investigator — St Georges University Hospitals
Locations (1):
- St Georges University Hospital, London, Tooting, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pegorie C, Liu B, Thilaganathan B, Bhide A. Ambulatory foetal ECG monitoring in low and high-risk pregnancies (AMBER2): a prospective cohort study protocol. BMJ Open. 2025 Sep 28;15(9):e096123. doi: 10.1136/bmjopen-2024-096123. PMID 41022451